CLINICAL TRIAL: NCT05716854
Title: Clinical ECG Study to Evaluate Electrophysiological Effects of Potential QT Prolonging Drugs With Novel ECG Biomarkers With Exposure-Response Analysis
Brief Title: Electrophysiological Effects of Potential QT Prolonging Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SCR-014
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Drug-induced QT Prolongation; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Clarithromycin; Pimozide; Moxifloxacin; Cobicistat

STUDY DESIGN:
Intervention Model Description: This clinical study consists of 2 parts: a 3-arm, 22-subject crossover study (Part 1) and a 4-arm, 22-subject crossover study (Part 2). These parts are included in the same protocol and study due to the similarity of the inclusion and exclusion criteria, similar procedures, and similar primary goals.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind, and the blind will be maintained through a randomization schedule held by the dispensing pharmacist. Treatments will be over-encapsulated. The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Part 1: Clarithromycin Administration Only (Active Comparator): Subjects in this arm will be administered Clarithromycin only over 3 days of dosing.
  Interventions: Drug: Clarithromycin
- Part 1: Pimozide Administration Only (Active Comparator): Subjects in this arm will be administered Pimozide only over 3 days of dosing.
  Interventions: Drug: Pimozide
- Part 1: Placebo (Placebo Comparator): Subjects in this arm will not be administered any drug. Will serve as placebo comparator arm.
  Interventions: Drug: Placebo (Part 1)
- Part 2: Moxifloxacin Administration Only (Active Comparator): Subjects in this arm will be administered Moxifloxacin only for 1 day of dosing.
  Interventions: Drug: Moxifloxacin
- Part 2: Cobicistat Administration Only (Active Comparator): Subjects in this arm will be administered Cobicistat only for 1 day of dosing.
  Interventions: Drug: Cobicistat
- Part 2: Moxifloxacin and Cobicistat Administration (Active Comparator): Subjects in this arm will be administered both Cobicistat and Moxifloxacin for 1 day of dosing.
  Interventions: Drug: Moxifloxacin and Cobicistat
- Part 2: Placebo (Placebo Comparator): Subjects in this arm will not be administered any drug. Will serve as placebo comparator arm.
  Interventions: Drug: Placebo (Part 2)

INTERVENTIONS:
Drug: Clarithromycin — Subjects receive the Clarithromycin intervention orally according to the following schedule:
  Day 1: 1 Clarithromycin 500 mg immediate release (IR) tablet twice (Clarithromycin 500 mg BID).
  Day 2: 2 Clarithromycin 500 mg immediate release (IR) tablets twice (Clarithromycin 1000 mg BID).
  Day 3: 2 Clarithromycin 500 mg immediate release (IR) tablets once (Clarithromycin 1000 mg QD).
  Other Names: Treatment A
  Arms: Part 1: Clarithromycin Administration Only
Drug: Pimozide — Subjects receive the Pimozide intervention orally according to the following schedule:
  Days 1-3: Pimozide 6 mg immediate release (IR) once per day.
  Other Names: Treatment B
  Arms: Part 1: Pimozide Administration Only
Drug: Placebo (Part 1) — Subjects receive matching placebo for treatments.
  Other Names: Treatment C
  Arms: Part 1: Placebo
Drug: Moxifloxacin — Subjects receive Moxifloxacin 800 mg orally once on day 1.
  Other Names: Treatment D
  Arms: Part 2: Moxifloxacin Administration Only
Drug: Cobicistat — Subjects receive Cobicistat 450 mg orally once on day 1.
  Other Names: Treatment E
  Arms: Part 2: Cobicistat Administration Only
Drug: Moxifloxacin and Cobicistat — Subjects receive Moxifloxacin 800 mg and Cobicistat 450 mg orally once on day 1.
  Other Names: Treatment F
  Arms: Part 2: Moxifloxacin and Cobicistat Administration
Drug: Placebo (Part 2) — Subjects receive matching placebo for treatments.
  Other Names: Treatment G
  Arms: Part 2: Placebo

SUMMARY:
Since 2005, FDA has required almost all new drugs be tested for their ability to prolong the QT interval through clinical studies. This requirement stems from the increased TdP risk QT interval prolongation can cause. However, the QT interval is an imperfect biomarker, as there are multiple drugs that can prolong the QT interval, without causing increased TdP occurrence. As such, numerous drugs labeled as causing QT prolongation, may in fact have no impact on TdP occurrence.

To address this problem, FDA, in collaboration with multiple external partners, has led an initiative to combine novel preclinical in vitro experiments within silico modeling and simulation followed by pharmacodynamic electrocardiographic (ECG) biomarkers. The goal is to use these novel computational and analytical tools to better predict TdP risk (beyond just the QT interval) by focusing on understanding the underlying mechanisms and applying an integrated biological systems approach.

This clinical study consists of 2 parts: a 3-arm, 22-subject crossover study (Part 1) and a 4-arm, 22-subject crossover study (Part 2). These parts are included in the same protocol and study due to the similarity of the inclusion and exclusion criteria, similar procedures, and similar primary goals.

DETAILED DESCRIPTION:
The risk of drug-induced Torsades de Pointes (TdP), a potentially fatal ventricular arrhythmia, has resulted in multiple drugs worldwide being removed from the market, as well as over 150 drugs being listed on CredibleMeds.org for QT prolongation or TdP association. In response, since 2005, FDA has required almost all new drugs be tested for their ability to prolong the QT interval through clinical studies. This requirement stems from the increased TdP risk QT interval prolongation can cause. However, the QT interval is an imperfect biomarker, as there are multiple drugs that can prolong the QT interval, without causing increased TdP occurrence. As such, numerous drugs labeled as causing QT prolongation, may in fact have no impact on TdP occurrence. While this labeling affects physician prescribing, it also has the potential to limit effective therapeutic options for patients.

To address this problem, FDA, in collaboration with multiple external partners, has led an initiative to combine novel preclinical in vitro experiments within silico modeling and simulation followed by pharmacodynamic electrocardiographic (ECG) biomarkers. The goal is to use these novel computational and analytical tools to better predict TdP risk (beyond just the QT interval) by focusing on understanding the underlying mechanisms and applying an integrated biological systems approach.

Recently, the International Council on Harmonization (ICH) released a new Guideline with updated Questions and Answers (Q&As) to the clinical (ICH E14) and nonclinical (ICH S7B) Guidelines for assessing the QT prolongation and proarrhythmic risk of non-antiarrhythmic drugs. The Q&A provides more guidance on the use of an integrated nonclinical analysis to support clinical QT assessment. This includes the comparison of the hERG safety margin of the investigational product to the safety margin of predominant hERG (the human Ether-à-go-go-Related Gene) blockers with a characterization of the concentration-QTc relationship based on a limited set of example drugs, i.e., ondansetron, moxifloxacin and dofetilide.

This clinical study consists of 2 parts: a 3-arm, 22-subject crossover study (Part 1) and a 4-arm, 22-subject crossover study (Part 2). These parts are included in the same protocol and study due to the similarity of the inclusion and exclusion criteria, similar procedures, and similar primary goals.

Part 1: Intermediate risk predominant hERG blocking drugs The FDA performed a literature review and identified 28 proarrhythmic drugs from available in vitro studies of cardiac ion channel IC50 (using HEK293 cells and the hERG 1a subunit). Two of these drugs, classified as intermediate risk "predominant hERG blocking" (pimozide and clarithromycin), have been identified as candidates for evaluation in Part 1. An aim of this study will be generating higher quality QT data on "intermediate risk" "predominant hERG" blocking drugs' effect on both electrocardiographic biomarkers, QTc and J-Tpeakc interval prolongation, at therapeutic and supratherapeutic exposures. These data will also be used to support assessment of the hERG safety margin threshold together with moxifloxacin, dofetilide, and ondansetron as described in the recently released ICH Q&A's.

Part 2: Combination of hERG and multi-ion channel block Part 2 of this study will assess the effects of a mixed ion channel blocking drug, cobicistat, on the QTc and J-Tpeakc interval alone and in combination with a predominant hERG blocking drug (moxifloxacin). Clinical data with cobicistat, a structural analog of ritonavir used as a pharmacokinetic enhancer in various anti-viral regimens, has demonstrated QTc shortening and PR prolongation with supratherapeutic doses. Whether this is a results of late sodium block, calcium channel block, or other features is unclear. Additional clinical data with cobicistat alone or in combination with moxifloxacin will enhance our understanding of the effects of mixed ion channel blocking on electrocardiographic biomarkers (QTc and J-Tpeakc interval).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an IRB approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy non-smoker who weighs at least 50 kg (110 lbs) and has a body mass index of 18.5 to 33.0 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, pulse oximetry, 12-lead ECG results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and check-in days.
5. Subject must test negative for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) by a rapid antigen test at check-in for all study periods.
6. Female subjects must be of non-childbearing potential (confirmed with follicle-stimulating hormone levels > 40 mIU/mL) or, if they are of childbearing potential, they must: 1) have negative serum HCG at screening and check-in 2) have been strictly abstinent for 1 month before check-in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1month after the last application of study drug; OR 3) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before check-in (Day -1) until at least 1 month after the end of the study.
7. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee) from at least 1 month before check-in (Day -1) until at least 3 months after the last dose of study drug.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Subject has a 12-lead safety ECG result at Screening or check-in (Day -1) with evidence of any of the following abnormalities:

   * QT corrected interval (QTc) using Fridericia correction (QTcF) >430 milliseconds (ms)
   * PR interval >220 ms or <120 ms
   * QRS duration >110 ms
   * Second- or third-degree atrioventricular block
   * Complete left or right bundle branch block or incomplete right bundle branch block
   * Heart rate <50 or >90 beats per minute
   * Pathological Q-waves (defined as Q wave >40 ms)
   * Ventricular pre-excitation
2. Subject has a history of unexplained syncope, structural heart disease, long QT syndrome, heart failure, myocardial infarction, angina, unexplained cardiac arrhythmia, torsade de pointes, ventricular tachycardia, or placement of a pacemaker or implantable defibrillator. Subjects shall also be excluded if there is a family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome.
3. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug. This includes prescription or nonprescription ophthalmic drugs. Note the only two drugs permitted are oral contraceptives and acetaminophen.
4. Subject is currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of dosing for this study.
5. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, electronic cigarettes) within 6 weeks of Screening. Subjects must refrain from using these throughout the study.
6. Subject has consumed alcohol, xanthine-containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 24 hrs of check-in. Subjects must refrain from ingesting these throughout the study.
7. Subject is unable to tolerate a controlled, quiet study conduct environment, including avoidance of music, television, movies, games, and activities that may cause excitement, emotional tension, or arousal during the prespecified time points (e.g., before and during ECG extraction windows).
8. Subject is unwilling to comply with study rules, including the study-specific diet, attempting to void at specified times (e.g., before ECG extraction windows), remaining quiet, awake, undistracted, motionless, and supine during specified times, and avoiding vigorous exercise as directed.
9. Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months before Screening, has a history of alcoholism or drug/chemical/substance abuse within 2 years before Screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits/hard liquor), or has a positive test result for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates) at Screening or Check-in of each period.
10. Subject has a history or evidence of a clinically significant disorder, condition, or disease (e.g., cancer, human immunodeficiency virus [HIV], hepatic or renal impairment) that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion. This includes subjects with any underlying medical conditions that the Investigator believes would put subjects at increased risk of severe illness from COVID-19 based on the Centers for Disease Control and Prevention (CDC) guidelines. The CDC lists cancer, chronic kidney disease, chronic obstructive pulmonary disease, immunocompromised state from solid organ transplant, severe obesity, serious heart conditions, sickle cell disease, pregnancy, smoking and type 2 diabetes mellitus as conditions that put subjects at increased risk. Additionally, the CDC lists asthma (moderate-to-severe), cerebrovascular disease, cystic fibrosis, hypertension, immunocompromised state or immune deficiencies, neurologic conditions such as dementia, liver disease, pulmonary fibrosis, thalassemia, BMI > 25.0, and type 1 diabetes mellitus as conditions that might put subjects at increased risk.
11. Subject has any signs or symptoms that are consistent with COVID-19 per CDC recommendations. These include subjects with fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea may have COVID-19. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
12. Subject has known or suspected allergies or sensitivities to the study drug.
13. Subject has a history of thoracic surgery.
14. Subject has any condition possibly affecting study drug absorption (e.g., gastrectomy, Crohn's disease, irritable bowel syndrome).
15. Subject has a skin condition likely to compromise ECG electrode placement.
16. Any individual with breast implants.
17. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at Screening or Check-In that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator. Tests may be repeated once for confirmation.
18. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
19. Subject has a mean systolic blood pressure <90 or >140 mmHg or a mean diastolic blood pressure <50 or >90 mmHg at either Screening or Check-in of Period 1.
20. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or is unlikely to complete the study due to poor venous access.
21. Female subject is currently pregnant or lactating or was within 3 months of the study.
22. Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days before Check-in of Period 1.
23. Subject has any other condition that precludes his or her participation in the study (as determined by the investigator).
24. Subject undergoes genetic testing for CYP2D6 phenotype and is a "poor metabolizer" (only for Part 1).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Plasma concentration of pimozide and clarithromycin associated with ΔΔQTc prolongation of 10 ms based on concentration-QTc analysis. | 1, 2, 2.5, 3, 4, 6, 8, 14, and 24 hours
Part 2: ΔΔJ-TpeakC between cobicistat and moxifloxacin compared to moxifloxacin based on ECG timepoint analysis. | -1, -0.5, 0 (pre-dose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 14, and 24 hours

SECONDARY OUTCOMES:
Part 1: ΔΔQTc for pimozide and clarithromycin at maximum drug concentration on day 3 based on concentration-QTc analysis. | 1, 2, 2.5, 3, 4, 6, 8, 14, and 24 hours
Part 1: ΔΔJ-TpeakC for pimozide and clarithromycin at maximum drug concentration on day 3 based on concentration-QTc analysis. | 1, 2, 2.5, 3, 4, 6, 8, 14, and 24 hours
Part 1: The margin (ratio) between hERG IC50 and free plasma concentration causing 10 ms QTc prolongation. | 1, 2, 2.5, 3, 4, 6, 8, 14, and 24 hours
Part 2: ΔΔQTc between cobicistat and moxifloxacin compared to moxifloxacin based on ECG timepoint analysis. | -1, -0.5, 0 (pre-dose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 14, and 24 hours
Part 2: ΔΔQTc for moxifloxacin, cobicistat, and moxifloxacin + cobicistat compared to placebo based on ECG timepoint analysis. | -1, -0.5, 0 (pre-dose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 14, and 24 hours
Part 2: ΔΔJ-Tpeakc for moxifloxacin, cobicistat, and moxifloxacin + cobicistat compared to placebo based on ECG timepoint analysis. | -1, -0.5, 0 (pre-dose), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 14, and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Boston, MSN, APNP, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as part of a manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as with any eventual publications.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Darpo B, Benson C, Dota C, Ferber G, Garnett C, Green CL, Jarugula V, Johannesen L, Keirns J, Krudys K, Liu J, Ortemann-Renon C, Riley S, Sarapa N, Smith B, Stoltz RR, Zhou M, Stockbridge N. Results from the IQ-CSRC prospective study support replacement of the thorough QT study by QT assessment in the early clinical phase. Clin Pharmacol Ther. 2015 Apr;97(4):326-35. doi: 10.1002/cpt.60. PMID 25670536
- [Background] Dutta S, Chang KC, Beattie KA, Sheng J, Tran PN, Wu WW, Wu M, Strauss DG, Colatsky T, Li Z. Optimization of an In silico Cardiac Cell Model for Proarrhythmia Risk Assessment. Front Physiol. 2017 Aug 23;8:616. doi: 10.3389/fphys.2017.00616. eCollection 2017. PMID 28878692
- [Background] Li Z, Ridder BJ, Han X, Wu WW, Sheng J, Tran PN, Wu M, Randolph A, Johnstone RH, Mirams GR, Kuryshev Y, Kramer J, Wu C, Crumb WJ Jr, Strauss DG. Assessment of an In Silico Mechanistic Model for Proarrhythmia Risk Prediction Under the CiPA Initiative. Clin Pharmacol Ther. 2019 Feb;105(2):466-475. doi: 10.1002/cpt.1184. Epub 2018 Aug 27. PMID 30151907
- [Background] Chang KC, Dutta S, Mirams GR, Beattie KA, Sheng J, Tran PN, Wu M, Wu WW, Colatsky T, Strauss DG, Li Z. Uncertainty Quantification Reveals the Importance of Data Variability and Experimental Design Considerations for in Silico Proarrhythmia Risk Assessment. Front Physiol. 2017 Nov 21;8:917. doi: 10.3389/fphys.2017.00917. eCollection 2017. PMID 29209226
- [Background] Li Z, Dutta S, Sheng J, Tran PN, Wu W, Chang K, Mdluli T, Strauss DG, Colatsky T. Improving the In Silico Assessment of Proarrhythmia Risk by Combining hERG (Human Ether-a-go-go-Related Gene) Channel-Drug Binding Kinetics and Multichannel Pharmacology. Circ Arrhythm Electrophysiol. 2017 Feb;10(2):e004628. doi: 10.1161/CIRCEP.116.004628. PMID 28202629
- [Background] Sager PT, Gintant G, Turner JR, Pettit S, Stockbridge N. Rechanneling the cardiac proarrhythmia safety paradigm: a meeting report from the Cardiac Safety Research Consortium. Am Heart J. 2014 Mar;167(3):292-300. doi: 10.1016/j.ahj.2013.11.004. Epub 2013 Dec 2. PMID 24576511
- [Background] McCreadie RG, Heykants JJ, Chalmers A, Anderson AM. Plasma pimozide profiles in chronic schizophrenics. Br J Clin Pharmacol. 1979 May;7(5):533-4. doi: 10.1111/j.1365-2125.1979.tb01001.x. No abstract available. PMID 475950
- [Background] Polis MA, Piscitelli SC, Vogel S, Witebsky FG, Conville PS, Petty B, Kovacs JA, Davey RT Jr, Walker RE, Falloon J, Metcalf JA, Craft C, Lane HC, Masur H. Clarithromycin lowers plasma zidovudine levels in persons with human immunodeficiency virus infection. Antimicrob Agents Chemother. 1997 Aug;41(8):1709-14. doi: 10.1128/AAC.41.8.1709. PMID 9257746
- [Background] Vance E, Watson-Bitar M, Gustavson L, Kazanjian P. Pharmacokinetics of clarithromycin and zidovudine in patients with AIDS. Antimicrob Agents Chemother. 1995 Jun;39(6):1355-60. doi: 10.1128/AAC.39.6.1355. PMID 7574530
- [Background] Darpo B, Benson C, Brown R, Dota C, Ferber G, Ferry J, Jarugula V, Keirns J, Ortemann-Renon C, Pham T, Riley S, Sarapa N, Ticktin M, Zareba W, Couderc JP. Evaluation of the Effect of 5 QT-Positive Drugs on the JTpeak Interval - An Analysis of ECGs From the IQ-CSRC Study. J Clin Pharmacol. 2020 Jan;60(1):125-139. doi: 10.1002/jcph.1502. Epub 2019 Aug 5. PMID 31378962
- [Background] Johannesen L, Vicente J, Mason JW, Erato C, Sanabria C, Waite-Labott K, Hong M, Lin J, Guo P, Mutlib A, Wang J, Crumb WJ, Blinova K, Chan D, Stohlman J, Florian J, Ugander M, Stockbridge N, Strauss DG. Late sodium current block for drug-induced long QT syndrome: Results from a prospective clinical trial. Clin Pharmacol Ther. 2016 Feb;99(2):214-23. doi: 10.1002/cpt.205. Epub 2015 Nov 28. PMID 26259627
- [Background] Mathias AA, German P, Murray BP, Wei L, Jain A, West S, Warren D, Hui J, Kearney BP. Pharmacokinetics and pharmacodynamics of GS-9350: a novel pharmacokinetic enhancer without anti-HIV activity. Clin Pharmacol Ther. 2010 Mar;87(3):322-9. doi: 10.1038/clpt.2009.228. Epub 2009 Dec 30. PMID 20043009
- [Background] Newman LM, Kankam M, Nakamura A, Conrad T, Mueller J, O'Donnell J, Osborn BL, Gu K, Saviolakis GA. Thorough QT Study To Evaluate the Effect of Zoliflodacin, a Novel Therapeutic for Gonorrhea, on Cardiac Repolarization in Healthy Adults. Antimicrob Agents Chemother. 2021 Nov 17;65(12):e0129221. doi: 10.1128/AAC.01292-21. Epub 2021 Oct 4. PMID 34606332
- [Background] Johannesen L, Vicente J, Gray RA, Galeotti L, Loring Z, Garnett CE, Florian J, Ugander M, Stockbridge N, Strauss DG. Improving the assessment of heart toxicity for all new drugs through translational regulatory science. Clin Pharmacol Ther. 2014 May;95(5):501-8. doi: 10.1038/clpt.2013.238. Epub 2013 Dec 12. PMID 24336137
- [Background] Holford NH, Coates PE, Guentert TW, Riegelman S, Sheiner LB. The effect of quinidine and its metabolites on the electrocardiogram and systolic time intervals: concentration--effect relationships. Br J Clin Pharmacol. 1981 Feb;11(2):187-95. doi: 10.1111/j.1365-2125.1981.tb01123.x. PMID 7213522
- [Background] Garnett C, Bonate PL, Dang Q, Ferber G, Huang D, Liu J, Mehrotra D, Riley S, Sager P, Tornoe C, Wang Y. Scientific white paper on concentration-QTc modeling. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):383-397. doi: 10.1007/s10928-017-9558-5. Epub 2017 Dec 5. PMID 29209907
- [Background] Vicente J, Simlund J, Johannesen L, Sundh F, Florian J, Ugander M, Wagner GS, Woosley RL, Strauss DG. Investigation of potential mechanisms of sex differences in quinidine-induced torsade de pointes risk. J Electrocardiol. 2015 Jul-Aug;48(4):533-8. doi: 10.1016/j.jelectrocard.2015.03.011. Epub 2015 Mar 12. PMID 25796102